CLINICAL TRIAL: NCT03748121
Title: Pranayama Assisted Psychotherapy in Patients With Post-traumatic Stress Disorder: a Randomized-controlled Trial
Brief Title: Yoga/Pranayama for Posttraumatic Stress Disorder
Acronym: YOGAPTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Heidemarie Haller, Postdoctoral Research Fellow, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-7703-BO
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Cognitive-Behavioral Therapy; Complementary Therapies; Yoga; Pranayama; Effectiveness; Safety; Randomized Controlled Trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and Therapists (Care Provider) could not be blinded according to the nature of the intervention. However, therapists will be blinded to allocation concealment as they do not be aware of the patients' group assignment at baseline assessment until they open the opaque randomization envelope, which contains the patient randomization number and group assignment. The random sequence generation and the envelopes were prepared by the study coordinator who is not involved patient recruitment. Patients received post intervention questionnaires from a study assistant/nurse of the respective outpatient department who is also blinded to the patients' group assignment. After completing the questionnaires, the study assistant will sent them to study coordinator so that the therapist could not influence the patients' answers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pranayama assisted Trauma-focused Cognitive Behavioral Therapy (TF-CBT) (Experimental): To prepare patients for the TF-CBT, they received 5-10 minutes of pranayama at the begin of each of the 10 TF-CBT units.
  Interventions: Behavioral: Pranayama assisted trauma-focused Cognitive Behavioral Therapy (TF-CBT)
- Trauma-focused Cognitive Behavioral Therapy (TF-CBT) (Active Comparator): Patients wait for 10 TF-CBT units and then are offered to learn pranayama.
  Interventions: Behavioral: Trauma-focused Cognitive Behavioral Therapy (TF-CBT)

INTERVENTIONS:
Behavioral: Pranayama assisted trauma-focused Cognitive Behavioral Therapy (TF-CBT) — The pranayama intervention is placed directly at the begin of the respective TF-CBT unit and will be repeated for 10 subsequent TF-CBT units. Pranayama contains the performance of Kapalabhati, Ujjayi, and/or Nadi Shodhana (for overall 1 minute) as well as following Kumbhaka (intentional respiratory reflex inhibition). Pranayama will be repeated 3 times before each TF-CBT unit.
  Arms: Pranayama assisted Trauma-focused Cognitive Behavioral Therapy (TF-CBT)
Behavioral: Trauma-focused Cognitive Behavioral Therapy (TF-CBT) — Trauma-focused Cognitive Behavioral Therapy (TF-CBT)
  Arms: Trauma-focused Cognitive Behavioral Therapy (TF-CBT)

SUMMARY:
This study aims to investigate the effect of a pranayama focused yoga intervention on post-traumatic symptom severity in patients with post-traumatic stress disorder undergoing standard psychotherapy/ trauma-focused cognitive-behavioral therapy (TF-CBT). Therefore, short pranayama sessions of 5-10 minutes will be provided to the patients directly at the begin of each of standard TF-CBT unit, while the control group will get standard TF-CBT alone. It should further be investigated, whether pranayama can enhance the affective tolerance of patients with post-traumatic stress disorder towards the used exposure techniques of TF-CBT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed PTSD according to ICD-10
* PCL-5 Score of at least 33 points
* Undergoing outpatient CBT
* Physical and mental ability to perform Pranayama

Exclusion Criteria:

* Severe comorbid mental or somatic disease that did not allow the patient to perform Pranayama
* Pregnancy
* Regular practice of Yoga or Pilates in the last 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Intensity of posttraumtic symptoms | week 10
  Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): The PCL-5 is a standard 20-item scale with a sum score ranging from 0 to 80 points. The cut-off point for clinically relevant symptom severity is 33 points.

SECONDARY OUTCOMES:
Health-related quality of life | week 10
  Short Form 12 Health Survey (SF-12): The SF-12 is a standard 12-item scale with two sum scores (physical and mental quality of life) ranging from 0 to 100 points.
Ability of social participation | week 10
  Patient-Reported Outcomes Measurement Information System - Ability to Participate in Social Roles and Activities Scale (PROMIS): The PROMIS-Social Participation Subscale is a standard 8-item scale ranging from 0 to 100 points with 100 points represent the highest possible ability to participate/function.
Anxiety | week 10
  Beck Anxiety Inventory (BAI): The BAI is a standard 21-items scale ranging from 0 to 63 points with 0-7 points = minimal anxiety, 8-15 points = mild anxiety, 16-25 points = moderate anxiety, and 26-63 points = clinically relevant anxiety.
Depression | week 10
  Beck Depression Inventory Revision (BDI-II): The BDI-II is a standard 21-items scale ranging from 0 to 63 points with 0-13 points =no/clinically not relevant depression/depression in remission, 14-19 points = mild depression, 20-28 points = moderate depression und 29-63 points = severe depression.
Distress Tolerance | week 10
  Distress Tolerance Scale (DTS): The DTS is a standard 15-item scale ranging from 0 to 75 points. Higher scores represent higher distress tolerance.
Emotion Regulation | week 10
  Emotion Regulation Scale (ERQ): The ERQ is a standard 10-item scale with 6 items are added to the Cognitive Reappraisal subscale ranging from 6 to 42 and 4 items are added to the Expressive Suppression subscale ranging from 4 to 28. Higher scores on the Cognitive Reappraisal subscale and lower ones on the Expressive Suppression subscale represent a better regulation of emotions.
Body Awareness | week 10
  Scale of Body Connection (SBC): The SBC is a standard 20-items scale ranging from 0 to 80 that contains two subscales: Body Awareness and Body Dissociation. Higher scores on Body Awareness and lower scores on Body Dissociation represent a better body awareness.
Breath Holding Duration | week 10
  Breath Holding Task (BHT): The BHT is standard test procedure for the measurement of ability of the suppression of the respiratory reflex. In PTSD patients, it is associated with distress tolerance.
Acute Emotional Stress | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10
  Emotional Stress Reaction Questionnaire (ESRQ): The ESRQ is standard 14-items scale ranging from -21 points (predominance of negative emotions) to +21 points (predominance of positive emotions). Patients received the ESRQ before and after each CBT unit.
Adverse Events | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10
  Number of patients with adverse events (and type of the adverse event)

OTHER OUTCOMES:
Treatment Expectation | week 0
  Treatment Credibility Scale (TCS): The TCS is a standard NRS scale ranging from 0 points (lowest expectation of treatment effectiveness) to 10 points (highest expectation of treatment effectiveness).

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof. MD, Study Director — University of Duisburg-Essen
Locations (1):
- Dietmar Mitzinger, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request.

REFERENCES:
- [Derived] Haller H, Mitzinger D, Cramer H. The integration of yoga breathing techniques in cognitive behavioral therapy for post-traumatic stress disorder: A pragmatic randomized controlled trial. Front Psychiatry. 2023 Apr 17;14:1101046. doi: 10.3389/fpsyt.2023.1101046. eCollection 2023. PMID 37139325